CLINICAL TRIAL: NCT07384468
Title: Ultrasound-Guided Stellate Ganglion Block Combined With Propofol for Perimenopausal Insomnia With Anxiety
Brief Title: Ultrasound-Guided Stellate Ganglion Block Plus Propofol for Perimenopausal Insomnia With Anxiety
Acronym: SGB-PROP-PIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaochen Ji (Other)
Responsible Party: Sponsor-Investigator, Xiaochen Ji, Principal Investigator, Cangzhou Central Hospital
Organization: Cangzhou Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZCH-SGB-PROP-INS-01
Record Dates: First submitted 2026-01-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Uterine Fibroids (UF)
Keywords: Stellate Ganglion Block; Laparoscopic Myomectomy; General Anesthesia; Perioperative Hemodynamics; Heart Rate Variability; Postoperative Recovery; Perioperative Stress Response; Postoperative Pain
MeSH Terms: conditions — Leiomyoma; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel assignment with two arms (ultrasound-guided right-sided stellate ganglion block plus standardized general anesthesia vs sham saline injection plus standardized general anesthesia).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors were blinded to group allocation. The anesthesiologist performing the stellate ganglion block was not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Block Group (Experimental): Patients received ultrasound-guided right-sided stellate ganglion block prior to anesthesia induction, followed by standardized general anesthesia for laparoscopic myomectomy.
  Interventions: Procedure: Ultrasound-Guided Stellate Ganglion Block
- General Anesthesia Group (Sham Comparator): Patients received an ultrasound-guided sham injection with an equal volume of normal saline at the stellate ganglion prior to anesthesia induction, followed by standardized general anesthesia for laparoscopic myomectomy.
  Interventions: Procedure: Sham Stellate Ganglion Block

INTERVENTIONS:
Procedure: Ultrasound-Guided Stellate Ganglion Block — Ultrasound-guided right-sided stellate ganglion block was performed prior to anesthesia induction. Using a high-frequency linear ultrasound probe at the C6 level, ropivacaine was injected into the prevertebral fascial plane between the longus colli muscle and prevertebral fascia.
  Arms: Combined Block Group
Procedure: Sham Stellate Ganglion Block — An ultrasound-guided sham procedure was performed prior to anesthesia induction, in which an equal volume of normal saline was injected at the same anatomical location without performing an active stellate ganglion block.
  Arms: General Anesthesia Group

SUMMARY:
Laparoscopic myomectomy is a commonly performed minimally invasive gynecologic procedure. However, surgical trauma, tracheal intubation, and pneumoperitoneum may induce pronounced perioperative stress responses, resulting in hemodynamic instability, postoperative pain, inflammatory activation, sleep disturbance, and anxiety, which can delay postoperative recovery.

Stellate ganglion block (SGB) is a sympathetic nerve modulation technique that has been shown to attenuate stress-related sympathetic overactivity. This study aimed to evaluate the clinical effects and safety of ultrasound-guided right-sided stellate ganglion block combined with standardized general anesthesia in patients undergoing laparoscopic myomectomy.

In this randomized controlled study, a total of 240 patients scheduled for laparoscopic myomectomy were randomly assigned to either a combined block group (ultrasound-guided right-sided SGB before anesthesia induction plus general anesthesia) or a general anesthesia group (sham saline injection plus general anesthesia). Perioperative hemodynamic parameters, heart rate variability, postoperative pain scores, analgesic requirements, recovery profiles, inflammatory stress markers, sleep quality, anxiety levels, and adverse events were compared between groups.

This study was retrospectively registered after completion. The results are intended to provide evidence for optimizing perioperative management and enhancing recovery in patients undergoing laparoscopic myomectomy.

DETAILED DESCRIPTION:
This single-center, randomized controlled clinical study was conducted to investigate the effects of ultrasound-guided right-sided stellate ganglion block (SGB) on perioperative stress responses and postoperative recovery in patients undergoing laparoscopic myomectomy under general anesthesia.

A total of 240 adult female patients scheduled for elective laparoscopic myomectomy were enrolled and randomly assigned in a 1:1 ratio to either the combined block group or the general anesthesia group. All participants received standardized general anesthesia with propofol-based induction and maintenance. In the combined block group, ultrasound-guided right-sided stellate ganglion block was performed prior to anesthesia induction using ropivacaine. In the control group, an identical ultrasound-guided procedure was conducted with injection of an equal volume of normal saline at the same anatomical location.

Perioperative management and postoperative analgesia protocols were standardized for both groups. Hemodynamic variables and heart rate variability parameters were recorded at predefined perioperative time points. Postoperative pain intensity was assessed using the visual analog scale, and analgesic consumption was recorded during the first 48 hours after surgery. Recovery indicators, including time to first flatus and ambulation, were documented. Inflammatory and stress-related biomarkers were measured preoperatively and at 24 hours postoperatively. Sleep quality and anxiety were evaluated using validated questionnaires before surgery and on postoperative day one. Adverse events were monitored and recorded throughout the perioperative period.

The study protocol was reviewed and approved by the Ethics Committee of Cangzhou Central Hospital (Approval No. 2024-332-03). Written informed consent was obtained from all participants prior to enrollment. The trial was retrospectively registered following study completion to enhance transparency and public accessibility of the study design and results.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 35 to 55 years.
* Diagnosed with uterine fibroids and scheduled for elective laparoscopic myomectomy.
* American Society of Anesthesiologists (ASA) physical status classification I or II.
* Normal cognitive function and ability to understand the study procedures.
* Provided written informed consent prior to participation.

Exclusion Criteria:

* Contraindications to stellate ganglion block, including coagulation disorders, infection at the puncture site, or allergy to local anesthetics.
* Severe dysfunction of major organs, including heart, liver, or kidney.
* Poorly controlled chronic diseases such as hypertension or diabetes mellitus.
* History of psychiatric disorders, chronic pain conditions, or long-term use of sedatives, analgesics, or medications affecting autonomic nervous system function.
* Preexisting significant sleep disorders prior to surgery.
* Abnormal cervical anatomy, history of cervical surgery, or radiotherapy.
* Anticipated difficult airway.
* Conversion to open surgery during the procedure.
* Failure of stellate ganglion block.
* Occurrence of serious adverse events related to the block procedure, such as nerve injury, arrhythmia, or local anesthetic systemic toxicity.
* Unplanned admission to the intensive care unit after surgery.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 233 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Mean Arterial Pressure During Airway Manipulation | Immediately after tracheal intubation and at extubation during surgery
  Mean arterial pressure (MAP), measured in mmHg.
Heart Rate During Airway Manipulation | Immediately after tracheal intubation and at extubation during surgery
  Heart rate (HR), measured in beats per minute.

SECONDARY OUTCOMES:
Low-Frequency (LF) Power of Heart Rate Variability | Pre-block (baseline), immediately after tracheal intubation, 5 minutes after pneumoperitoneum creation, at the end of surgery, and at extubation
  Low-frequency (LF) power of heart rate variability, measured in ms²/Hz.
Low-Frequency/High-Frequency (LF/HF) Ratio of Heart Rate Variability | Pre-block (baseline), immediately after tracheal intubation, 5 minutes after pneumoperitoneum creation, at the end of surgery, and at extubation
  Low-frequency to high-frequency (LF/HF) ratio of heart rate variability.
Postoperative Pain Intensity at Rest | 6 hours, 12 hours, and 24 hours after surgery
  Pain intensity assessed using the Visual Analog Scale (VAS), scored from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating more severe pain.
Postoperative Patient-Controlled Intravenous Analgesia (PCIA) Use | Within 48 hours after surgery
  Number of patient-controlled intravenous analgesia (PCIA) pump button presses.
Use of Rescue Analgesia | Within 48 hours after surgery
  Proportion of participants receiving rescue analgesia.
Time to First Flatus | From end of surgery to first postoperative flatus (assessed up to hospital discharge, up to 7 days)
  Time from completion of surgery to first postoperative flatus, measured in hours.
Time to First Ambulation | From end of surgery to first postoperative ambulation (assessed up to hospital discharge, up to 7 days)
  Time from completion of surgery to first postoperative ambulation, measured in hours.
Length of Hospital Stay | From completion of surgery to hospital discharge (up to 7 days)
  Total length of postoperative hospital stay, measured in days.
Serum Interleukin-6 Level | Baseline (pre-intervention) and 24 hours after surgery
  Serum interleukin-6 (IL-6) concentration.
Serum Cortisol Level | Baseline (pre-intervention) and 24 hours after surgery
  Serum cortisol concentration.
Serum Norepinephrine Level | Baseline (pre-intervention) and 24 hours after surgery
  Serum norepinephrine concentration.
Sleep Quality | Preoperatively and postoperative day 1
  Sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI), with total scores ranging from 0 to 21, where higher scores indicate poorer sleep quality.
Anxiety Level | Preoperatively and postoperative day 1
  Anxiety assessed using the Self-Rating Anxiety Scale (SAS), with standard scores ranging from 20 to 80, where higher scores indicate greater anxiety severity.
Adverse Events | Within 48 hours after surgery
  Incidence of postoperative adverse events, including nausea and vomiting, dizziness, headache, and shoulder pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Cangzhou Central Hospital, Cangzhou, Hebei, China

IPD SHARING:
Plan to Share IPD: No